CLINICAL TRIAL: NCT00897897
Title: Clinical Trial Protocol for Therapeutic MRI-guided High Intensity Focused Ultrasound Ablation of Uterine Fibroids
Brief Title: Therapeutic Magnetic Resonance Imaging (MRI)-Guided High Intensity Focused Ultrasound (HIFU) Ablation of Uterine Fibroids
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Philips Healthcare (Industry)
Collaborators: Philips Medical Systems (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 996233
Record Dates: First submitted 2009-05-11; First posted 2009-05-12 (Estimated); Results first posted 2011-11-11 (Estimated); Last update posted 2012-12-04 (Estimated); Status verified 2012-12

CONDITIONS: Uterine Fibroids
Keywords: Uterine Leiomyomas; Fibroids; HIFU; Ablation; High Intensity Focused Ultrasound
MeSH Terms: conditions — Leiomyoma; Myofibroma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treated leiomyomas (Other): Pre- or peri-menopausal women with symptomatic uterine fibroids who desire a uterine sparing procedure receive a treatment with the Philips MRI-guided HIFU system. Patients must have completed child bearing prior to enrolling in this study.
  Interventions: Device: Philips MRI-guided HIFU system

INTERVENTIONS:
Device: Philips MRI-guided HIFU system — HIFU is the use of focused ultrasound energy to penetrate through soft tissue and causes localized high temperatures (55°C to 70°C) for a few seconds within the target producing well defined regions of protein denaturation, irreversible cell damage, and coagulative necrosis.
  Other Names: Sonalleve

SUMMARY:
This study is to confirm the safety and technical effectiveness of MRI guided High Intensity Focused Ultrasound (HIFU) in ablating uterine tissue associated with symptomatic leiomyomas. The importance of this therapy is that it offers a non-invasive, uterine sparing procedure for the treatment of uterine fibroids in pre- and peri- menopausal women.

MRI guided high intensity focused ultrasound uses ultrasound to heat and thermally ablate fibroid tissue. The MRI system identifies the ultrasound path and monitors heat rise in the fibroid tissue. The goal of the study is to show treatment safety and technical effectiveness. MR-guided HIFU will be performed in patients who pass inclusion/exclusion criteria. Safety, quality of life, and imaging endpoints will be evaluated in all study patients.

The goal of this study is to demonstrate that:

1. The safety profile is acceptable (safety)
2. Actual MR-HIFU ablated volumes (as measured with contrast enhanced MRI) match the intended volumes (technical effectiveness)
3. When intended, volumes greater than 20% of the fibroid volume can be successfully ablated (technical effectiveness)

The investigators' hypothesis is that greater than 70% of fibroids will have concordance between intended lesion volume and actual lesion volume while maintaining an acceptable safety profile.

DETAILED DESCRIPTION:
Fibroids occur in 20-50% of women over 30 years of age, and with increasing size produce pain, menorrhagia, pressure, bloating and urinary and bowel compression symptoms. Fibroids may also cause infertility. Uterine leiomyomas are benign tumors originating from smooth muscle cells of the uterus and occasionally the smooth muscle of uterine blood vessels. Fibroids are estrogen dependent tumors ranging in size and number and can be found within the myometrium(intramural), at the uterine periphery extending to the serosa (subserosal), or pushing into the uterine cavity (submucosal). Symptomatic fibroids impact health and well-being of the female including lost work hours and reduced quality of life.

Current medical treatments include invasive removal of the fibroid (hysterectomy, myomectomy), drug therapy (GnRH analogues or progestin compounds) or treatments causing necrosis of the fibroid tissue such as ablation (freezing or heating) or embolization. For the relief of symptoms, women wishing to preserve the uterus may choose between invasive procedures of myomectomy, Uterine Artery Embolization (UAE), ablation or cryotherapy. The surgically invasive procedures require anesthesia, hospital stays, and long recovery periods. HIFU may offer an alternative to the above mentioned surgically invasive procedures.

In MRI-guided High Intensity Focused Ultrasound (HIFU), the ultrasound generated by the transducer is focused into a small focal tissue volume at specific target locations. During treatment, the beam of focused ultrasound energy penetrates through soft tissue and causes localized high temperatures (55°C to 70°C) for a few seconds within the target producing well defined regions of protein denaturation, irreversible cell damage, and coagulative necrosis. The MRI system allows 3D planning, means of measuring the temperature increase generated by HIFU, and the capability to quantifying the energy/dose delivered to the treatment zone.

This study is a multi-center, single arm, non-randomized trial evaluating the safety, technical effectiveness and volume treatment capabilities of the Philips MR-guided HIFU system in the treatment of symptomatic uterine fibroid patients. Patients who have symptomatic uterine fibroids, who are eligible according to the inclusion and exclusion criteria and provide informed consent will be enrolled in this study. It is anticipated that women will participate in the study for a 2month period to include the screening, HIFU treatment and post treatment follow-up.

This clinical study is designed to confirm safety and demonstrate technical effectiveness of the Philips HIFU system for Uterine Fibroid treatment. Safety will be primarily assessed by evaluating minor complications and adverse events, and technical effectiveness will primarily be assessed with MRI measurements. Specific primary and secondary endpoints are detailed below.

The study will use a combination of three primary endpoints: MR imaging of ablated volumes and minor complications/adverse events analysis to establish the safety and technical effectiveness of the Philips MR-HIFU system. These endpoints will determine the trial success.

The treatment capabilities and technical effectiveness of the Philips MR-guided HIFU system will be assessed by (measurement type is noted in parentheses)

1. Comparing the actual MR-measured ablated volumes to MR thermal dose predicted volumes

   Safety of the Philips MR-guided HIFU system will be demonstrated by
2. Evaluating any minor complications or adverse events that result from the MR-guided HIFU treatment
3. Verifying with MR imaging that no unintended lesions are formed as a result of the Treatment

   Our hypothesis is that greater than 70% of fibroids will have concordance between intended lesion volume and actual lesion volume while maintaining an acceptable safety profile.

   In addition, the following endpoints will be collected to supplement the primary outcomes:
4. Pain and discomfort scores before, during and after treatment: These endpoints will be recorded using a 10-point visual analog scale for pain 4-point scale for discomfort.
5. Return to Activity: This duration in days will be determined by the time after which the patients return to work (i.e. days after leaving the hospital) or to the usual activities for those not employed.
6. Length of Hospital Stay (LOS): This duration in hours will be measured from the time the patient will arrive to the hospital until she will leave the hospital.
7. Quality of Life questionnaires: the SF-36(http://www.sf36.org/tools/SF36.shtml) and UFS-QoL (which includes SSS)

ELIGIBILITY:
Inclusion Criteria:

* Women, age between 18 and 59 years
* Weight < 140kg
* Pre- or peri-menopausal
* Uterine size < 24 weeks
* Transformed SSS score > 40
* Normal Cervical cell assessment by PAP
* Symptomatic Fibroid disease
* Dominant fibroid greater than or equal to 3cm and less than or equal to 12 cm

Exclusion Criteria:

* Other Pelvic Disease
* Desire for future pregnancy
* Significant systemic disease even if controlled
* Positive pregnancy test
* Hematocrit < 25%
* Scarring or other interference of the HIFU beam
* MRI or contrast contraindicated
* Fibroids not quantifiable on MRI
* Calcifications around or throughout uterine tissues
* Communication barrier

Ages: 18 Years to 59 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2009-04; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Herve Trillaud, Prof, MD, Principal Investigator — Hospital St. Andre, Bordeaux, France; Lim Hyo Keun, MD, Principal Investigator — Samsung Medical Center, Seoul, Korea; Willem Mali, Prof, MD, Principal Investigator — University Medical Center - Utrecht, Netherlands; Joerg Barkhausen, Prof, MD, Principal Investigator — University Hospital Schleswig-Holstein, Lübeck, Germany
Locations (4):
- Hospital St. Andre, Bordeaux, France
- University Hospital Schleswig-Holstein, Lübeck, Germany
- University Medical Center, Utrecht, Netherlands
- Samsung Medical Center, Seoul, South Korea

REFERENCES:
- [Background] Spies JB, Coyne K, Guaou Guaou N, Boyle D, Skyrnarz-Murphy K, Gonzalves SM. The UFS-QOL, a new disease-specific symptom and health-related quality of life questionnaire for leiomyomata. Obstet Gynecol. 2002 Feb;99(2):290-300. doi: 10.1016/s0029-7844(01)01702-1. PMID 11814511
- [Background] Stewart EA, Gedroyc WM, Tempany CM, Quade BJ, Inbar Y, Ehrenstein T, Shushan A, Hindley JT, Goldin RD, David M, Sklair M, Rabinovici J. Focused ultrasound treatment of uterine fibroid tumors: safety and feasibility of a noninvasive thermoablative technique. Am J Obstet Gynecol. 2003 Jul;189(1):48-54. doi: 10.1067/mob.2003.345. PMID 12861137
- [Background] Hindley J, Gedroyc WM, Regan L, Stewart E, Tempany C, Hynyen K, Mcdannold N, Inbar Y, Itzchak Y, Rabinovici J, Kim HS, Geschwind JF, Hesley G, Gostout B, Ehrenstein T, Hengst S, Sklair-Levy M, Shushan A, Jolesz F. MRI guidance of focused ultrasound therapy of uterine fibroids: early results. AJR Am J Roentgenol. 2004 Dec;183(6):1713-9. doi: 10.2214/ajr.183.6.01831713. PMID 15547216
- [Background] Leon-Villapalos J, Kaniorou-Larai M, Dziewulski P. Full thickness abdominal burn following magnetic resonance guided focused ultrasound therapy. Burns. 2005 Dec;31(8):1054-5. doi: 10.1016/j.burns.2005.04.019. Epub 2005 Jun 20. No abstract available. PMID 15970389
- [Background] Fennessy FM, Tempany CM. MRI-guided focused ultrasound surgery of uterine leiomyomas. Acad Radiol. 2005 Sep;12(9):1158-66. doi: 10.1016/j.acra.2005.05.018. PMID 16099686
- [Background] Stewart EA, Rabinovici J, Tempany CM, Inbar Y, Regan L, Gostout B, Hesley G, Kim HS, Hengst S, Gedroyc WM. Clinical outcomes of focused ultrasound surgery for the treatment of uterine fibroids. Fertil Steril. 2006 Jan;85(1):22-9. doi: 10.1016/j.fertnstert.2005.04.072. PMID 16412721
- [Background] Fennessy FM, Tempany CM, McDannold NJ, So MJ, Hesley G, Gostout B, Kim HS, Holland GA, Sarti DA, Hynynen K, Jolesz FA, Stewart EA. Uterine leiomyomas: MR imaging-guided focused ultrasound surgery--results of different treatment protocols. Radiology. 2007 Jun;243(3):885-93. doi: 10.1148/radiol.2433060267. Epub 2007 Apr 19. PMID 17446521
- [Background] Mara M, Fucikova Z, Maskova J, Kuzel D, Haakova L. Uterine fibroid embolization versus myomectomy in women wishing to preserve fertility: preliminary results of a randomized controlled trial. Eur J Obstet Gynecol Reprod Biol. 2006 Jun 1;126(2):226-33. doi: 10.1016/j.ejogrb.2005.10.008. Epub 2005 Nov 15. PMID 16293363

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment was initiated on March 19, 2009 and completed on April 24, 2010.
Groups:
- Treated Leiomyomas: Pre- or peri-menopausal women with symptomatic uterine fibroids who desire a uterine sparing procedure. Patients must have completed child bearing prior to enrolling in this study.
  Patients underwent a single Magnetic Resonanc Imaging-guided High Intensity Focused Ultrasound (MR-HIFU) therapy session as an outpatient procedure, and were followed up for 30 days following treatment.
Period: Overall Study
Arm/Group | Treated Leiomyomas
Started | 33
Completed | 33
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treated Leiomyomas
Number analyzed (Participants) | 33
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 33
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 44.8 (5.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33
  Male | 0
Region of Enrollment [Number; unit: participants]
  France | 16
  Germany | 4
  Netherlands | 3
  Korea, Republic of | 10

OUTCOME MEASURES:

1. Primary Outcome: Adverse Events/Subject Resulting From HIFU Treatment of the Uterine Fibroids
Description: The number of Adverse Events reported during the study, divided by the total number of treated subjects. This corresponds to the mean number of Adverse Events per subject.
Time Frame: 30 days after treatment
Measure: Mean (Standard Deviation); unit: Adverse Event/subject
Arm/Group | Treated Leiomyomas
Number analyzed (Participants) | 33
Adverse Event/subject | 2.6 (2.6)

2. Secondary Outcome: Fibroid Symptom Severity Score (SSS) From the Uterine Fibroid Symptoms - Quality of Life (UFS-QoL) Questionnaire.
Description: Mean absolute change in the Symptom Severity Score (SSS) of the Uterine Fibroid Symptoms - Quality of Life (UFS-QoL) questionnaire after fibroid treatment with HIFU.
  The SSS is a scale from 0-100, where 0 corresponds to no symptoms and 100 corresponds to the most severe symptoms.
Time Frame: At baseline and at 30 days following treatment
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Treated Leiomyomas
Number analyzed (Participants) | 33
scores on a scale | -13.6 (17.7)

ADVERSE EVENTS:
Time Frame: Adverse Event information was collected from baseline to 30 days after treatment, i.e. 30 days
Arm/Group | Treated Leiomyomas
Serious Adverse Events (participants affected / at risk) | 0/33
Other Adverse Events (participants affected / at risk) | 23/33
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treated Leiomyomas (N=33)
Abdominal Pain (General disorders) | 10 (10) — Abdominal pain such as cramping, pain or tenderness
Back Pain (General disorders) | 4 (4)
Bloating (General disorders) | 4 (4)
Fatigue and Tiredness (General disorders) | 6 (6)
Headache (General disorders) | 3 (3)
Nausea (General disorders) | 2 (2)
Vaginal Bleeding (General disorders) | 2 (2)
Urinary Burning (General disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less